CLINICAL TRIAL: NCT07152470
Title: An Open Label 100 Person Study Evaluating a Natural Supplement for Weight Loss and Fat Loss in a Real World Setting.
Brief Title: An Open Label 100 Person Study Evaluating a Natural Supplement for Weight Loss and Fat Loss.
Status: Active, not recruiting | Type: Observational
Sponsor: Prostasis, LLC, dba Tonum Health (Industry)
Responsible Party: Sponsor
Other Study IDs: Motus1001
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy Diet with Daily Exercise (>4 days per week): Participants consumed a strict healthy diet and daily exercise (>30 mins) as determined by nutritionists who were randomly assigned to participants to review their wellness tracker and conduct periodic 1:1 coaching sessions
  Interventions: Behavioral: Diet and Exercise Tracking
- Average Diet with Moderate Exercise (2-3 days per week): Participants consumed an average diet with 2-3 days of exercise per week (>30 mins) as determined by nutritionists who were randomly assigned to participants to review their wellness tracker and conduct periodic 1:1 coaching sessions
  Interventions: Behavioral: Diet and Exercise Tracking
- Average Diet with No Exercise (0 days per week): Participants consumed an average diet with zero days of exercise per week as determined by nutritionists who were randomly assigned to participants to review their wellness tracker and conduct periodic 1:1 coaching sessions
  Interventions: Behavioral: Diet and Exercise Tracking
- Poor Diet with No Exercise (0 days per week): Participants consumed a poor diet with zero days of exercise per week as determined by nutritionists who were randomly assigned to participants to review their wellness tracker and conduct periodic 1:1 coaching sessions
  Interventions: Behavioral: Diet and Exercise Tracking

INTERVENTIONS:
Behavioral: Diet and Exercise Tracking — To determine if diet and/or exercise had any impact on weight loss while taking motus.

SUMMARY:
The goal of this clinical trial is to learn if motus, a natural supplement can support healthy weight loss and fat loss in a real world setting without caloric restrictions or exercise requirements.

The main questions it aims to answer are:

Can a daily dose of motus result in statistically significant weight loss over 3 month and 6 month time points.

Participants will:

Weigh-in at baseline and every week thereafter Take drug motus every day Complete a food tracker app for every meal and drink product consumed daily Complete an exercise tracker for any activities performed daily Complete weekly satisfaction surveys on various topics

DETAILED DESCRIPTION:
A prospective, observational human study was conducted with 100 participants (ages 25-68, BMI ≥25) over an initial 12-week period, followed by a 12-week extension phase for 40 continuing participants. All subjects received motus (4-capsule daily dose) and were instructed to track food intake and exercise via food tracker app and digital fat measurement scales. No caloric restriction was mandated, and participants could optionally receive nutritional counseling. Weekly weigh-ins and quality of life surveys were completed. No financial compensation was provided. Participants were stratified post hoc into three behavioral groups based on food and activity logs reviewed by registered dietitians: Category 1 (healthy diet + exercise 4+ times per week), Category 2 (average diet + exercise 2-3 times per week), Category 3 (average diet + no exercise) and Category 4 (poor diet + no exercise).

ELIGIBILITY:
Inclusion Criteria:

* BMI >25
* Willing to complete daily diary and weekly weigh-ins
* Willing to take motus daily

Exclusion Criteria:

* BMI<25
* Unwilling to complete daily diary and weekly weigh-ins
* Currently taking a prescribed weight loss medication
* Currently or planning to be pregnant

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 patients in the United states
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Total Weight Loss | 26 weeks
  Total weight loss as a percentage of total body weight
Body Fat Loss | 26 weeks
  Total body fat loss compared to lean mass loss

CONTACTS AND LOCATIONS:
Locations (1):
- Tonum Health, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided